CLINICAL TRIAL: NCT02326701
Title: RV Function by Strain and MRI
Brief Title: RV Function Evaluation Assessed by Strain and Validated by MRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: DG001-HMO-CTIL
Record Dates: First submitted 2014-11-02; First posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-10

CONDITIONS: Right Ventricular Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Echocardiographic assessment of right ventricular function is an important diagnostic tool, and is a challenge due to the unique structure and anatomy of the right ventricle. Lately a new technique has been developed and used for evaluating both the left and the right ventricle function. This technique, called two dimensional (2D) speckle tracking, is based on detecting speckles in the myocardial tissue and using them as acoustic markers. The movement of these speckles represents the movement of the tissue, and allows us to evaluate its function, contraction and relaxation, this by calculating the strain rate, which is the speed of the speckles, and the strain, which is the distance between them.

In the last few years this technique has been used to evaluate the systolic function of the right ventricle in several pathological conditions, such as pulmonary hypertension, pulmonary embolism and amyloidosis. Nonetheless, so far there has been little data on the normal RV strain and strain rate values.

In this study the investigators aim to validate two dimensional (2D) speckle tracking measurements of the RV function by comparing them to strain measurements by cardiac MRI. Each patient performing cardiac MRI for any indication will perform an echocardiography examination in addition, and strain analysis performed on the cardiac MRI will be compared with two dimensional speckle tracking analysis performed on the echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Age: More than 18

Exclusion Criteria:

* Age: Children
* Unconcious patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients performing MRI for any indication
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of 2D Echo and Echo strain measurements versus MRI measurements | 1 year
  RV dimensions, RV function, RV strain measurements compared to MRI measurements

SECONDARY OUTCOMES:
Rehospitalization | 2 years
  Time from index event to timing and length of rehospitalization (based on hospital data and completed with phone interview when necessary)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel